CLINICAL TRIAL: NCT07330089
Title: Retention of Pits and Fissure Sealants on Non Carious vs Initial Carious Enamel Lesions in Posterior Teeth, a Non Randomized Clinical Study
Brief Title: Retention of Pits and Fissure Sealants on Non Carious vs Initial Carious Enamel Lesions in Posterior Teeth
Status: Not yet recruiting | Type: Observational
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Shoaib Rahim, Associate Professor, Foundation University Islamabad
Other Study IDs: FUCDOP2512
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Dental Enamel; Dental Enamel Hypomineralization; Dental Enamel Hypoplasia
Keywords: pit and fissure sealants; pit sealant; fissure sealant
MeSH Terms: conditions — Dental Enamel Hypomineralization; Dental Enamel Hypoplasia; Van der Woude syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: pit and fissure sealant non carious enamel lesions (ICDAS score 0): pits and fissure sealants will be applied in non carious (sound) enamel surfaces of posterior permanent teeth and the retention will the evaluated at 3, 6 , and 12 months.
- Group 2: pit and fissure sealant on Initial caries enamel lesions (ICDAS I and II): pits and fissure sealants will be applied in initial carious enamel surfaces of posterior permanent teeth and the retention will the evaluated at 3, 6 , and 12 months.

SUMMARY:
This clinical study is planned to be conducted to compare retention rates of pits and fissure sealants on non carious (ICDAS score 0) vs Initial carious enamel lesions (ICDAS Score 1,2) in posterior permeant teeth at 3 months, 6 months and 12 months follow-up. This will help us guide follow-up strategies for optimal caries prevention.

DETAILED DESCRIPTION:
It is an observational, non randomized quasi experimental study design in which patients aged between 7 to 18years will be selected for the study. After obtaining informed consent, the 1st permanent molars and 2nd permanent molar (if erupted) will be evaluated for carious ICDAS SCORE. On the basis of score, the participants will be divided into two groups i.e. non carious group and initial carious group. sample size of 210 teeth will be allocated in each group. Irrespective of the carious status either non carious or initial caries enamel lesions, tooth surfaces will be etched with 37% phosphoric acid (total etch Ivoclar Vivadent) for 15 seconds till frosty white appearance is achieved. the molars will then be sealed by Conseal F sealant and light cured for 20 seconds. The patients will then be called on follow-up at 3, 6 and 12 months and retention of the sealants will be checked using Simonson criteria with the help of explorer. Simonson score I - Completely retained sealants, score II- partially retained sealants , score III complete loss of sealants. All this information will be added in the clinical Performa. After this data collection , data will be analyzed using SPSS 26.0. to compare the proportion of sealants that were lost will be compared using chi square test and p value of 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Fully erupted maxillary and mandibular 1st and 2nd molars with antagonist teeth present.
* ICDAS score 0,I,II
* Age 7 to 18 years
* Both genders included

Exclusion Criteria:

* permanent teeth requiring restorations,
* uncooperative patients
* patients unwilling for follow-ups
* molars withy antagonist teeth not present
* mentally and physically handicapped patients
* patients with parafunctional habits
* patients undergoing orthodontic treatments

Ages: 7 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients reporting to Paedodontics and Operative dentistry department of FUCD&H will be selected according to inclusion criteria after history, clinical examination.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
retention of pit and fissure sealant on non carious vs initial carious enamel lesions- 12 months follow-up study. | from January 2026 to June 2027
  retention of pit and fissure sealants will be accessed through simonsen's criteria on non carious (210 teeth) vs initial carious enamel (210 teeth) with 12 month follow-up to guide follow-up strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Fizza Sherazi, BDS, Principal Investigator — Foundation University Islamabad

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vitamins to protect against and reverse aging. Dermatol Nurs. 2002 Jun;14(3):206-7. No abstract available. PMID 12099072
- [Background] McKenna G. A clinical guide to advanced minimum intervention restorative dentistry (1st ed). Br Dent J. 2024 Dec;237(11):834. doi: 10.1038/s41415-024-8183-0. No abstract available. PMID 39672849
- [Background] Demineralization and remineralization dynamics and dental caries.
- [Background] Evaluating the effectiveness of dental sealants in caries prevention and tooth protection
- [Background] Banerjee A, Splieth C, Breschi L, Fontana M, Paris S, Burrow M, Crombie F, Foster Page L, Gaton-Hernandez P, Giacaman RA, Gugnani N, Hickel R, A Jordan R, Leal S, Lo E, Tassery H, Thomson WM, Manton DJ, Schwendicke F. When to intervene in the caries process? A Delphi consensus statement. Br Dent J. 2020 Oct;229(7):474-482. doi: 10.1038/s41415-020-2220-4. PMID 33037372
- [Background] Microscopic evaluation of fissure patterns of posterior permanent teeth: An in vitro study
- [Background] Pit and Fissure Sealants as a Viable Preventive Tool for Dental Caries
- [Background] Beresescu L, Pacurar M, Bica CI, Vlasa A, Stoica OE, Dako T, Petcu B, Esian D. The Assessment of Sealants' Effectiveness in Arresting Non-Cavitated Caries Lesion-A 24-Month Follow-Up. Healthcare (Basel). 2022 Aug 30;10(9):1651. doi: 10.3390/healthcare10091651. PMID 36141263
- [Background] Carrillo Ortiz AE, Olvera Fuentes CA, Garcia Perez A, Rodriguez Chavez JA, Villanueva Gutierrez T, Flores Ruiz HM, Mora Navarrete KA. Prevalence and severity of dental caries using ICDAS in predicting treatment needs in Mexican school-age children. J Clin Pediatr Dent. 2024 Nov;48(6):144-151. doi: 10.22514/jocpd.2024.134. Epub 2024 Nov 3. PMID 39543891
- Available data/document: literature review — https://www.dental-research.com/idr/article/view/403 — esearchgate.net/publication/377562421_Pit_and_Fissure_Sealants_as_a_Viable_Preventive_Tool_for_Dental_Caries